CLINICAL TRIAL: NCT07080086
Title: The Effect of Preoperative Biological Age on Intraoperative Hemodynamics and Postoperative Renal Function
Brief Title: The Effect of Preoperative Biological Age on Hemodynamics and Renal Function
Status: Completed | Type: Observational
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: KY-20240924-09
Record Dates: First submitted 2025-07-15; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2023-09

CONDITIONS: Acute Kidney Injury; Acute Kidney Disease; Intraoperative Hypotension; Post-induction Hypotension
Keywords: Intraoperative Hypotension; post-induction hypotension; Acute Kidney Injury; Acute kidney disease; Biological age; Biological aging
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Biological age: PhenoAge and Klemera-Doubal method biological age (KDM-BA), were utilized. PhenoAge was calculated using the combination of chronological age and nine clinical biomarkers (albumin, SCr, glucose, C-reactive protein (CRP), lymphocyte percentage, mean cell volume (MCV), red blood cell distribution width (RDW), alkaline phosphatase, and white blood cell count (WBC)). KDM-BA was calculated by chronological age and nine clinical biomarkers (albumin, SCr, CRP, alkaline phosphatase, systolic blood pressure, blood urea nitrogen, forced expiratory volume in one second (FEV1), glycated haemoglobin, and total cholesterol).

SUMMARY:
Background The aim of this study is to explore the potential value of preoperative biological age as a predictor of intraoperative hemodynamic changes and postoperative renal function injury.

Methods Collect data using medical record system and surgical anesthesia system, and gather patients who have undergone surgery. Calculate the preoperative biological age of the patient and analyze the correlation between preoperative biological age accelerated aging and intraoperative hemodynamics and postoperative renal function damage.

DETAILED DESCRIPTION:
With the intensification of population aging, the number of patients undergoing surgical procedures has been increasing year by year. However, traditional age indicators cannot fully reflect the physiological condition and surgical risks of patients. In clinical practice, preoperative evaluation is usually based on the patient's actual age, but this method fails to fully consider individual biological differences. As a new evaluation indicator, biological age can more accurately reflect an individual's physiological status and health level by comprehensively considering multiple biomarkers. Therefore, biological age has gradually become one of the important parameters for predicting surgical risk. The stability of intraoperative hemodynamics is crucial for the prognosis of surgical patients. Research has shown that intraoperative blood pressure fluctuations, heart rate variability, and other hemodynamic abnormalities are closely related to the occurrence of postoperative complications. Postoperative renal dysfunction (AKI) is a common and serious postoperative complication, especially more common in elderly patients. Previous studies have found that the occurrence of AKI is not only related to intraoperative hemodynamic disorders, but also significantly influenced by the patient's underlying health status. However, current research on the impact of biological age on intraoperative hemodynamics and its relationship with postoperative renal function injury is still limited. Further exploration of the relationship between preoperative biological age and intraoperative hemodynamic parameters, as well as their predictive value for postoperative renal function injury, will help improve the accuracy of preoperative risk assessment, optimize intraoperative management strategies, and ultimately improve patients' postoperative prognosis. Therefore, this study aims to provide a new predictive tool for clinical practice and a basis for personalized surgical management by systematically evaluating the impact of biological age on intraoperative hemodynamics and postoperative renal function injury.

Based on hospital data, evaluate the hemodynamic fluctuations and incidence of postoperative renal function damage in patients of different biological ages undergoing high-risk surgery. The study aims to verify whether biological age can be independent of traditional clinical evaluation indicators, provide more accurate prediction of perioperative risks for patients, and provide scientific basis for individualized treatment decision-making.

ELIGIBILITY:
Inclusion Criteria:

* Surgical pateints

Exclusion Criteria:

* (1) Lacking valid demographic information; (2) Lacking valid biological age; (3) Lacking blood pressure records

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing surgery with complete anaesthetic records
Sampling Method: Non-Probability Sample
Enrollment: 268833 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
The incidence ofn AKI | Within 7 days postoperative,
  Pateints encompasses an escalation in SCr of 50% or more, an increment of at least 0.3 mg/dL within 48 hours, or the need for RRT including haemodialysis, peritoneal dialysis, continuous renal replacement therapy, and kidney transplant. It was based on the 2012 Kidney Disease: Improving Global Outcomes (KDIGO) guidelines.
The incidence of AKD | Within 8-90 days post-surgery
  AKD was defined by a surge in SCr by more than 50%, or the initiation of RRT such as haemodialysis, peritoneal dialysis or continuous RRT.
The incidence of IOH | During intraoperative period
  IOH was defined as the presence of intraoperative epoque with MAP below 60 mmHg.
The incidence of PIH | From induction of general anesthesia to 20 minutes post-induction.
  PIH was defined as at least one measurement of SAP below 90 mmHg.

SECONDARY OUTCOMES:
The incidence of AKI 2+ | 0-7 days post-surgery
  AKI 2+ was identified as an elevation in SCr to a level at least twice that of the baseline measurement.
Cumulative duration of IOH and PIH | During surgery
  Calculate the cumulative duration below the threshold value
The cumulative AUC of IOH and PIH. | During surgery
  Total area under each threshold (areas under the curve (AUC) measured in mmHg*minutes).

CONTACTS AND LOCATIONS:
Overall Officials: Yali Ge, MD, Study Director — The First Affiliated Hospital with Nanjing Medical University

IPD SHARING:
Plan to Share IPD: No